CLINICAL TRIAL: NCT00197977
Title: Addressing Patients' Expectations of Total Knee Arthroplasty: Developing and Testing an Educational Intervention in a Randomized Trial
Brief Title: Addressing Patients' Expectations of Total Knee Arthroplasty in a Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 98101
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Knee Osteoarthritis; Arthroplasty, Replacement, Knee
Keywords: knee arthritis; total knee arthroplasty; expectations; education
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Educational program to address patients' expectations

SUMMARY:
The goals of this study are to develop and test an educational intervention to address patients' expectations of long-term outcomes of total knee arthroplasty.

DETAILED DESCRIPTION:
The first goal of this study is to develop an educational intervention to address patients' expectations of long-term outcomes of total knee arthroplasty. The intervention will be structured according to the expectations listed in the Hospital for Special Surgery Total Knee Replacement Expectations Survey. The second goal is to test the intervention in a randomized trial. An additional goal is to compare patients' self-reported knee symptoms with radiographic findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for this study if they are 40 years of age or older and are scheduled for primary total knee arthroplasty at the Hospital for Special Surgery.

Exclusion Criteria:

* Patients will be excluded from this study for the following reasons: if they are not fluent in English; if they are not going to attend the preoperative knee replacement class; if they are unable to complete the surveys; if they refuse to participate.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2001-11; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the within-patient change between pre and post program scores measured by the Hospital for Special Surgery Total Knee Replacement Expectations Survey.

SECONDARY OUTCOMES:
The secondary outcome is to compare patient-reported symptoms with radiographic ratings of disease activity.
The secondary outcome is to determine if expectations after the class coincide more closely with orthopedic surgeons expectations

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Mancuso, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Mancuso CA, Sculco TP, Wickiewicz TL, Jones EC, Robbins L, Warren RF, Williams-Russo P. Patients' expectations of knee surgery. J Bone Joint Surg Am. 2001 Jul;83(7):1005-12. doi: 10.2106/00004623-200107000-00005. PMID 11451969
- [Background] Mancuso CA, Ranawat CS, Esdaile JM, Johanson NA, Charlson ME. Indications for total hip and total knee arthroplasties. Results of orthopaedic surveys. J Arthroplasty. 1996 Jan;11(1):34-46. doi: 10.1016/s0883-5403(96)80159-8. PMID 8676117
- [Background] Blake VA, Allegrante JP, Robbins L, Mancuso CA, Peterson MG, Esdaile JM, Paget SA, Charlson ME. Racial differences in social network experience and perceptions of benefit of arthritis treatments among New York City Medicare beneficiaries with self-reported hip and knee pain. Arthritis Rheum. 2002 Aug;47(4):366-71. doi: 10.1002/art.10538. PMID 12209481
- [Background] Peterson MG, Hollenberg JP, Szatrowski TP, Johanson NA, Mancuso CA, Charlson ME. Geographic variations in the rates of elective total hip and knee arthroplasties among Medicare beneficiaries in the United States. J Bone Joint Surg Am. 1992 Dec;74(10):1530-9. PMID 1469013
- [Result] Mancuso CA, Graziano S, Briskie LM, Peterson MG, Pellicci PM, Salvati EA, Sculco TP. Randomized trials to modify patients' preoperative expectations of hip and knee arthroplasties. Clin Orthop Relat Res. 2008 Feb;466(2):424-31. doi: 10.1007/s11999-007-0052-z. Epub 2008 Jan 10. PMID 18196427